CLINICAL TRIAL: NCT02264652
Title: High Definition Cathodal Transcranial Direct Current Stimulation for Treatment of Refractory Partial Onset Epilepsy
Acronym: HD-TDCS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00622
Record Dates: First submitted 2014-10-01; First posted 2014-10-15 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy
Keywords: Refractory; Partial; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HD Transcranial Direct Stimulation (Experimental): Genuine cathodal HD-tDCS approximately 2mA will be delivered through High-Definition electrodes that will be arranged on the skull according to a 4x1-ring configuration with the central cathodal electrode placed over the identified target and surrounding return electrodes forming approximately a 5-cm radius ring.
  Interventions: Device: HD Transcranial Direct Stimulation

INTERVENTIONS:
Device: HD Transcranial Direct Stimulation — Genuine cathodal HD-tDCS will be delivered through High Definition electrodes that will be arranged on the skull according to a 4x1 ring configuration.
  Other Names: HD-tDCS

SUMMARY:
High-Definition transcranial Direct Current Stimulation (HD tDCS)

Genuine cathodal HD-tDCS will be delivered through High-Definition electrodes that will be arranged on the skull according to a 4x1-ring configuration with the central cathodal electrode placed over the identified target and surrounding return electrodes forming approximately a 5-cm radius ring.

Aim: To explore whether a novel form of tDCS can be a safe noninvasive treatment that could potentially suppress seizures in refractory partial-onset epilepsy.

DETAILED DESCRIPTION:
1 Introduction This document is a protocol for a human research study. This study is to be conducted in accordance with US government research regulations, and applicable international standards of Good Clinical Practice, and institutional research policies and procedures.

1.1 Background Focal Status epilepticus (FSE) is characterized by a prolonged, self-sustaining, and anatomically discrete seizures that last longer than one hour (at times as long as days or weeks) and that are associated with a definable neurologic behavior (Schomer 2005). Symptoms in FSE can vary according to the function of the brain area affected, can vary in discharge, and can be as simple as a repetitive limb movement as seen in epilepsy partialis continua (EPC), or as subtle as an inability to write a command or name an object. Prevalence of EPC is estimated to be 1 per one million (Cockerell 1996). A large proportion of FSE episodes are resultant from acute neurologic insult such as stroke or hemorrhage, although, at times, the cause of FSE remains unknown. FSE treatment should commence promptly upon its recognition using predefined treatment protocols. The goal of treatment is the rapid termination of the seizure to minimize the acute and chronic effects of this emergency and to allow for the prompt assessment and management of the underlying precipitant (Loddenkemper 2011).

Furthermore, patients may suffer from refractory partial onset epilepsy, and suffer from frequent seizures despite maximizing medical therapy, which may place them at higher risk of having FSE or EPC.

Yet many instances of FSE, EPC, and refractory partial onset epilepsy which is resistant to pharmacotherapy, and require nonpharmacologic treatment.

Accordingly, the investigatorspropose a Phase-1 clinical trial to test the safety and tolerability of High Definition Transcranial Direct Current Stimulation (HD-tDCS), a -noninvasive technology with the capacity to suppress seizures in patients with frequent partial onset seizures, and eventually FSE or EPC. The investigators plan to use the Soterix HD-tDCS device. The device is a current-controlled source which generates a constant output current. In other words, the device automatically maintains constant output current by decreasing or increasing the output voltage needed as long as it does not surpass device compliance voltage, which provides an added safety measure.

The HD-tDCS device poses a non-significant risk because

1. The device is not an implant with potential for serious risk to health, safety, or welfare of subject
2. The device is not purported for use supporting or sustaining human life with potential for serious risk to health safety or welfare of subject
3. The device is not for substantial use in diagnosing, curing, mitigating, or treating disease or otherwise preventing impairment of human health with a potential for serious risk to health safety or welfare of subject
4. The device does not otherwise present a serious risk to the health safety or welfare of a subject.

The investigators anticipate that this will be a step toward eventual wider application of HD-tDCS.

tDCS Basics: tDCS is a painless and safe method for focal brain stimulation. tDCS is based on decades-old observations that neuronal firing is modulated by low amplitude electrical direct current (DC). Specifically, when applied to the cerebral cortex, cathodal DC inhibits neuronal firing. The mechanisms by which cathodal DC reduces neuronal firing likely relate to hyper-polarization of the soma membrane which occurs when the apical dendrites neuron are oriented toward the cathode in a constant electric field. The practical application of tDCS is simple: low amplitude DC is administered via broad scalp electrodes (typically saline-saturated sponges) such that the cerebral cortex is exposed to cathodal DC beneath one of the electrodes - the remaining, (anodal) electrodes can be placed anywhere else on the body, or as proposed below, circumferentially around the cathode. tDCS methods have also recently been adapted to rats for experimental work with disease models (Rotenberg 2008; Kabakov 2012). Over 600 studies have been published using standard tDCS without significant adverse events. In a recently published safety and tolerability study on 131 subjects involved in tDCS experiments at the University of Pennsylvania. no significant adverse events occurred. With commonly reported mild side effects of tingling (76%), itching (68%), burning (54%), and pain (25%). Direct electrical current stimulation is presently FDA-approved for extracranial use, FDA applications for cranial stimulation (tDCS) for management of mood disorder and chronic pain is in progress. Currently, there have been a number of clinical protocols using tDCS for cranial applications (including previous approved protocols of the PI), which have considered tDCS a non-significant or minimal risk device (please see attached documentation).

Figure 1: Principle of tDCS induced reduction in excitability. (left) Cathodal tDCS results in outward directed cortical current, which hyperpolarizes somatic cell membranes. This in turn, reduces excitability. Anodal has opposite effects. HD-tDCS technology allows uni-directional polarization (cathodal/reduced excitability only) as well as stimulation of a small cortical target. Thus, while leveraging the well-established mechanisms of DC control and safety of tDCS, HD-tDCS allows us to explore, for the first time, targeted hyperpolarization for seizure control. (right) As established over decades of research (on right panel from Purpura and McMurty, 1965) DC current instantly modulates neuronal firing in a direction specific manner with cathodal stimulation suppressing firing, as well as epileptiform activity (below).

tDCS Advantages: tDCS units are inexpensive and light-weight. The electrical supply can be derived from conventional 9-volt batteries. The scalp electrodes can be fastened in seconds. tDCS can be combined easily with other therapies, such as those that may be required for resuscitation of an acutely-injured patient. tDCS is presently under investigation as a treatment for epilepsy, where excess cortical excitability is a prominent feature of the disease process, and where neuronal inhibition may be beneficial. Thus for SE, tDCS may offer a practical therapeutic option analogous to hypothermia or pharmacologic suppression of neuronal activity but with the benefit of easy, rapid and focal application in the setting of acute seizure or other form of brain injury.

Figure 2: Soterix Medical Inc. (SMI) HD-tDCS system including battery powered base unit, HD electrodes, and cap. The system has been validated in clinical trials and designated non-significant-risk by the FDA. SMI develops custom HD electrodes and "cups" which can be designed to integrate into EEG head-gear. The EASYcap headgear is shown with 4x1 HD electrode montage. Using the 10/20 system for electrode recording (filled circle) allows interlaced site for positioning of HD electrodes (open circles). The EASYcap provides for a range of adult and pediatric sizes. The system is portable, can be deployed simply, and even be integrated with EEG or used while the subject is moving.

1.2 Preclinical Data Recent clinical studies of cathodal tDCS that focused on chronic treatment of epilepsy show a mild anti-epileptic effect when tDCS is delivered interictally. The rationale behind interictal tDCS application is the reliance on the tDCS effects that outlast stimulation (plasticity). Though results from early animal and clinical studies suggest that such a plasticity-based approach warrants further consideration, here, the investigators propose to exploit the well-established acute effects of DC currents. Thus, what is mechanistically innovative in our approach is leveraging the robust acute effect of DC polarization (Durand 2001; Kabakov 2012). Refractory partial onset epilepsy represents a sustained state of brain hyper-excitability (analogous to slice models), which is expected to be instantly suppressed by weak DC.

High definition transcranial direct current stimulation (HD-tDCS) has an established safety and tolerability profile and is entering into the clinical arena for treatment of a number of neurologic disease states, such as mood disorder and chronic pain, and post-stroke motor deficit, where patients may benefit from focal modulation of cortical excitability. There has been similar tolerability data in a small number of subjects for HD-tDCS (Minhas 2010). Some subjects may experience skin irritation or redness after treatment that resolves within hours. However, in our hands at 1mA per HD electrodes, lasting skin irritations (>24h) have never been observed (N>100) even in prolonged studies (N>40). Many patients who have received both standard and HD-tDCS treatments report less sensations from HD-tDCS, likely because the electrolyte gel produces better contact with the skin compared to saline-soaked pads (Kuo et al). Indeed a NSR designation for the proposed study was obtained by the FDA (please see supporting documents)..

Recent studies by our group and others have extended tDCS experiments to preclinical experiments in rat seizure models, and demonstrated that electrical control with tDCS aborts ongoing seizures and reduces associated brain injury. Here the investigators propose to apply cathodal HD-tDCS (Fig 2), the inhibitory variant of this technology, specifically to suppress cortical excitability and terminate seizures in a well-selected group of patients who demonstrate frequent focal onset seizures.

Figure 3: Comparison of neuromodulation focality using the HD-tDCS 4x1-Ring deployment vs. conventional tDCS (left) High-resolution individualized finite element model FEM computer simulations. (top) Conventional tDCS with large "sponge" pad electrodes results in diffuse and un-focal brain stimulation, which is bi-directional (both depolarized/activated and hyperpolarized/inhibited regions). (bottom) In contrast, HD-tDCS Ring stimulation results in highly targeted cortical area stimulation. Directly under the electrodes this is unidirectional (hyperpolarization only). These improvements achieved with HD-tDCS are highly relevant to the clinical aims of this proposal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9 to 65 years
2. Focal-onset neocortical epilepsy (as determined by semiology, EEG, and/or MRI)
3. Frequent (>50% of EEG record) focal epileptiform discharges on EEG and/or frequent (defined as average of ≥2 daily seizures) focal-onset clinical seizure, refractory to medical anti-epileptic treatment. For the purposes of this study, any patient who has been treated with three or more AEDs at therapeutic doses for at least four weeks per drug will be considered medically refractory.
4. Seizure onset must be localizable by clinical semiology, EEG or MRI.
5. Subjects or guardians must be competent to sign an informed consent indicating awareness of the investigational nature of this study, treatment, benefits and procedures involved.

Exclusion Criteria:

1. Age over 65 years or under 9 years.
2. Implanted cardiac pacemakers, cochlear implants, implanted medication pump, or intracardiac line.
3. Within past six months, history of active heart disease, stroke, respiratory disease, or increased intracranial pressure such as after infarction or trauma.
4. Pregnant women. A urine test will be conducted on all post-menarchal females of childbearing age and potential to verify they are not pregnant.
5. History of significant head trauma (loss of consciousness >10 minutes) within the past 6 months.
6. Currently taking tricyclic anti-depressants, bupropion, or neuroleptic medications.
7. Intracranial metal (e.g., cortical stimulator, deep brain stimulator, intraventricular catheter) within 4 cm of optimal stimulation site. Location of cranial metal (e.g. skull screws) should be carefully documented.
8. Neurodegenerative disease.
9. Radiographic or electrophysiologic evidence for deep structure seizure focus (e.g., mesial temporal sclerosis or periventricular heterotopia)
10. Inability to remain seated and relatively still for 30 minutes.
11. Benign rolandic epilepsy.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
EEG monitoring | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Boston Children's Hospital - Neurology, Boston, Massachusetts
  - Neurology, New York, New York